CLINICAL TRIAL: NCT03102229
Title: Real-time Activity Monitoring to Prevent Admissions During RadioTherapy
Acronym: RAMPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Nitin Ohri, Associate Professor, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-6398
Record Dates: First submitted 2017-01-23; First posted 2017-04-05 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Cancer of the Head and Neck; Cancer of Lung; Cancer of Esophagus; Cancer of Stomach
Keywords: Activity Monitoring; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activity Monitoring (Experimental): 1. Enhanced Supportive Care - Status Checks Would occur everyday during treatment when a patient is deemed high-risk based on activity level. Other Names: •Daily Status Checks
  2. Enhanced Supportive Care - Referrals On an as-need basis, high risk patients can be referred to our nutritionist or palliative care doctor. Other Names: •Referrals
  Interventions: Other: Enhanced Supportive Care - Status Checks; Other: Enhanced Supportive Care - Referrals

INTERVENTIONS:
Other: Enhanced Supportive Care - Status Checks — Would occur everyday during treatment when a patient is deemed high-risk.
  Other Names: Daily Status Checks
Other: Enhanced Supportive Care - Referrals — On an as-need basis, high risk patients can be referred to our nutritionist or palliative care doctor.
  Other Names: Referrals

SUMMARY:
This study will aim to demonstrate that implementation of a rapid, multidisciplinary supportive care program for patients receiving chemoradiotherapy who are deemed to be at high risk for hospitalization based on real-time pedometer data will reduce the rate of hospitalization during chemoradiotherapy or within four weeks of radiotherapy completion.

DETAILED DESCRIPTION:
Primary Objective

* To demonstrate that implementation of a rapid, multidisciplinary supportive care program for patients receiving chemoradiotherapy who are deemed to be at high risk for hospitalization based on real-time pedometer data will reduce the rate of hospitalization during chemoradiotherapy or within four weeks of radiotherapy completion.

Secondary Objectives

* To demonstrate the feasibility of a program of rapid, multidisciplinary supportive care triggered by real-time pedometer data.
* To characterize the interventions enacted by our multidisciplinary supportive care team.
* To explore if interventions enacted by our multidisciplinary team for patients with low recent step counts lead to increased step counts in subsequent weeks compared to historical controls.
* To collect biospecimens for future correlative studies examining associations between blood/urine biomarkers and patient activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ECOG performance status 0-2
* Able to ambulate independently (without the assistance of a cane or walker)
* Diagnosis of invasive malignancy of the head and neck region, lung, esophagus, or stomach
* Planned treatment with fractionated (≥15 treatments) external beam radiotherapy with concurrent chemotherapy (or cetuximab) with curative intent (including preoperative or postoperative treatment)
* Women of childbearing potential must:

  * Have a negative serum or urine pregnancy test within 72 hours prior to the start of study therapy
  * Agree to utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study therapy is completed
  * Be advised of the importance of avoiding pregnancy during trial participation and the potential risks of an unintentional pregnancy
* All patients must sign study specific informed consent prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients hospitalized during treatment or within 4 weeks after completing radiotherapy. | During chemoradiotherapy or within 4 weeks after completion of radiotherapy.
  The primary endpoint of this study is hospitalization during chemoradiotherapy or within 4 weeks after completion of radiotherapy.

SECONDARY OUTCOMES:
Activation of the enhanced supportive care protocol | During chemoradiotherapy or within 4 weeks after completion of radiotherapy.
  Activation of the enhanced supportive care protocol (multidisciplinary evaluation and daily nursing/physician visits) based on recent step count data.
Frequency of clinician visits and supportive care measures implemented. | During chemoradiotherapy or within 4 weeks after completion of radiotherapy
  Clinician visits and supportive care measures that result from activation of the enhanced supportive care protocol
Patient-reported quality of life scores | During chemoradiotherapy or within 4 weeks after completion of radiotherapy.
  Patient-reported quality of life scores, measured using the EORTC QLC-C30 questionnaire.
Treatment-related toxicities | During chemoradiotherapy or within 4 weeks after completion of radiotherapy.
  Treatment-related toxicities, scored using CTCAE version 4.03.
Disease status | During chemoradiotherapy and up to two years after completion of radiotherapy.
  Disease progression or recurrence
Survival status | During chemoradiotherapy and and up to two years after completion of radiotherapy.
Modified Glasgow Prognostic Score | From time of registration to up to 4 weeks after completion of radiotherapy.
  Modified Glasgow Prognostic Score will be measured as a function of the C-Reactive Protein and Albumin levels that are collected throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No